CLINICAL TRIAL: NCT02532686
Title: DAAOI-2 add-on Treatment for Treatment-resistant Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsien-Yuan Lane, Department of Psychiatry, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSC-101-2314-B-039-030-MY3
Record Dates: First submitted 2015-08-10; First posted 2015-08-26 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia
Keywords: Treatment resistant; DAAOI; NMDA
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAAOI-2 (Experimental): DAAOI-2: 500-2000mg/d
  Interventions: Drug: DAAOI-2
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DAAOI-2 — 500-2000mg/d, oral, for 6 weeks
  Arms: DAAOI-2
Drug: placebo — oral, for 6 weeks
  Arms: placebo

SUMMARY:
Pharmacotherapy for schizophrenia has limitations such as residual positive and negative symptoms, cognitive deficits and intolerable side effects. Refractory schizophrenia is still a difficult clinical issue at present. According to the N-methyl-D-aspartate (NMDA) hypothesis, adjuvant NMDA-enhancing agents may have therapeutic benefit. DAAOI-2, a D-amino acid oxidase (DAAO) inhibitor, is a NMDA-enhancing agent. The aim of this project is to examine the effectiveness and safety of DAAOI-2 add-on treatment for treatment-resistant schizophrenia patients in a randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Pharmacotherapy for schizophrenia has limitations such as residual positive and negative symptoms, cognitive deficits and intolerable side effects. Refractory schizophrenia is still a difficult clinical issue at present. According to the N-methyl-D-aspartate (NMDA) hypothesis, many clinical trials on NMDA-enhancing agents were studied. Adjuvant NMDA-enhancing agents, including glycine, D-amino acids such as D-serine, and sarcosine (a glycine transporter I inhibitor), revealed beneficial but limited efficacy for positive and negative symptoms.

The aim of this project is to examine the effectiveness and safety of DAAOI-2 add-on treatment for treatment resistant schizophrenia patients in a randomized, double-blind, placebo - controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the DSM-IV criteria of schizophrenia
* Treatment resistant: No satisfactory response to at least two kinds of antipsychotics
* Remain symptomatic but without clinically significant fluctuation and the antipsychotic doses are unchanged for at least 3 months
* Have a minimum baseline total score of 70 on the Positive and Negative Syndrome Scale (PANSS)
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Meet DSM-IV criteria of substance (including alcohol) abuse or dependence
* Meet DSM-IV criteria of mental retardation
* Serious medical or neurological illness
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale(PANSS) | baseline
Positive and Negative Syndrome Scale(PANSS) | 2 weeks after the trial
Positive and Negative Syndrome Scale(PANSS) | 4 weeks after the trial
Positive and Negative Syndrome Scale(PANSS) | 6 weeks after the trial (The end of the trial)
Assessment of Negative symptoms(SANS) | baseline
Assessment of Negative symptoms(SANS) | 2 weeks after the trial
Assessment of Negative symptoms(SANS) | 4 weeks after the trial
Assessment of Negative symptoms(SANS) | 6 weeks after the trial (The end of the trial)

SECONDARY OUTCOMES:
PANSS subscales | baseline
PANSS subscales | 2 weeks after the trial
PANSS subscales | 4 weeks after the trial
PANSS subscales | 6 weeks after the trial (The end of the trial)
Clinical Global Impression (CGI) | baseline
Clinical Global Impression (CGI) | 2 weeks after the trial
Clinical Global Impression (CGI) | 4 weeks after the trial
Clinical Global Impression (CGI) | 6 weeks after the trial (The end of the trial)
Global assessment of function (GAF) | baseline
Global assessment of function (GAF) | 2 weeks after the trial
Global assessment of function (GAF) | 4 weeks after the trial
Global assessment of function (GAF) | 6 weeks after the trial (The end of the trial)
Hamilton Depression Rating Scale (HAMD) | baseline
Hamilton Depression Rating Scale (HAMD) | 2 weeks after the trial
Hamilton Depression Rating Scale (HAMD) | 4 weeks after the trial
Hamilton Depression Rating Scale (HAMD) | 6 weeks after the trial (The end of the trial)
Quality of life scale (QOL) | baseline
Quality of life scale (QOL) | 2 weeks after the trial
Quality of life scale (QOL) | 4 weeks after the trial
Quality of life scale (QOL) | 6 weeks after the trial (The end of the trial)
"Measurement and Treatment Research to Improve Cognition in Schizophrenia [MATRICS] | baseline
  An intergrated score from 7 domains:
  1. speed of processing: category fluency, trail making A, and digit symbol - coding from Wechsler adult intelligence scale (WAIS-III);
  2. sustained attention: continuous performance test;
  3. verbal and nonverbal working memory: backward digit span and spatial span from Wechsler memory scale (WMS-III);
  4. verbal learning and memory: word listing from WMS-III;
  5. visual learning and memory: visual reproduction from WMS-III;
  6. reasoning and problem solving: maze from Wechsler intelligence scale for children (WISC-III);
  7. social cognition: the managing emotions branch of Mayer-Salovey-Caruso emotional intelligence test (MSCEIT)
"Measurement and Treatment Research to Improve Cognition in Schizophrenia [MATRICS] | 6 weeks after the trial (The end of the trial)
  An intergrated score from 7 domains:
  1. speed of processing: category fluency, trail making A, and digit symbol - coding from Wechsler adult intelligence scale (WAIS-III);
  2. sustained attention: continuous performance test;
  3. verbal and nonverbal working memory: backward digit span and spatial span from Wechsler memory scale (WMS-III);
  4. verbal learning and memory: word listing from WMS-III;
  5. visual learning and memory: visual reproduction from WMS-III;
  6. reasoning and problem solving: maze from Wechsler intelligence scale for children (WISC-III);
  7. social cognition: the managing emotions branch of Mayer-Salovey-Caruso emotional intelligence test (MSCEIT)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan